CLINICAL TRIAL: NCT01709513
Title: A Randomized, Double-Blind, Double-Dummy, Active-Controlled Study to Evaluate the Efficacy and Safety of REGN727/SAR236553 in Patients With Primary Hypercholesterolemia Who Are Intolerant to Statins
Brief Title: Study of Alirocumab (REGN727/SAR236553) in Patients With Primary Hypercholesterolemia and Moderate, High, or Very High Cardiovascular (CV) Risk, Who Are Intolerant to Statins (ODYSSEY ALTERNATIVE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R727-CL-1119
Record Dates: First submitted 2012-10-08; First posted 2012-10-18 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Ezetimibe; alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Atorvastatin (statin rechallenge arm) (Other): Atorvastatin 20 mg over-encapsulated tablets orally once daily (QD) for 24 weeks and placebo (for alirocumab) subcutaneous (SC) injection every two weeks (Q2W) for 24 weeks added to stable lipid-modifying therapy (LMT).
  Interventions: Drug: Atorvastatin; Drug: Placebo
- Ezetimibe (Active Comparator): Ezetimibe 10 mg over-encapsulated tablets orally QD for 24 weeks and placebo (for alirocumab) SC injection Q2W for 24 weeks added to stable LMT.
  Interventions: Drug: Ezetimibe; Drug: Placebo
- Alirocumab 75 mg/ up to 150 mg (Experimental): Alirocumab 75 mg SC injection Q2W for 24 weeks and placebo (for atorvastatin/ezetimibe) over-encapsulated tablets orally QD for 24 weeks added to stable LMT. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on cardiovascular risk.
  Interventions: Drug: Alirocumab; Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin over-encapsulated tablets.
  Arms: Atorvastatin (statin rechallenge arm)
Drug: Ezetimibe — Ezetimibe over-encapsulated tablet.
  Other Names: Zetia
  Arms: Ezetimibe
Drug: Alirocumab — Alirocumab SC injection of 1 mL into the abdomen, thigh, or outer area of the upper arm.
  Other Names: REGN727/SAR236553
  Arms: Alirocumab 75 mg/ up to 150 mg
Drug: Placebo — Placebo for alirocumab, ezitimibe and atorvastatin.

SUMMARY:
This is a randomized, double-blind, double-dummy, active-controlled, parallel-group, multi-national, multi-center study to compare alirocumab (REGN727/SAR236553) versus ezetimibe in participants with primary hypercholesterolemia and moderate, high, or very high CV risk, who are intolerant to statins. An atorvastatin arm is added to determine that the population selected in the study is a truly statin intolerant population by assessing skeletal muscle-related adverse events.

ELIGIBILITY:
Inclusion:

1. Patients with primary hypercholesterolemia [Heterozygous Familial Hypercholesterolemia (heFH) or non-FH] with moderate, high or very high CV risk and a history of statin intolerance
2. Provide signed informed consent

Exclusion:

1. Calculated serum LDL-C <70 mg/dL (1.81 mmol/L) and very high CV risk at the screening visit
2. Calculated serum LDL-C <100 mg/dL (2.59 mmol/L) and high or moderate CV risk at the screening visit
3. A 10-year fatal cardiovascular disease risk score <1% at the screening visit

(The inclusion/ exclusion criteria provided above is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2012-09-30 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (70):
- United States (41):
  - Anaheim, California
  - Beverly Hills, California
  - Mission Viejo, California
  - Newport Beach, California
  - Northridge, California
  - Thousand Oaks, California
  - Hartford, Connecticut
  - Boynton Beach, Florida
  - Jacksonville, Florida
  - Lakeland, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Trinity, Florida
  - Addison, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Auburn, Maine
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - Clifton, New Jersey
  - New York, New York
  - Poughkeepsie, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Marion, Ohio
  - Danville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Port Matilda, Pennsylvania
  - Scranton, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Summerville, South Carolina
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
- Austria (3):
  - Feldkirch
  - Graz
  - Innsbruck
- Canada (3):
  - Chicoutimi, Quebec
  - Montreal (2 Locations), Quebec
  - Sainte-Foy, Quebec
- France (6):
  - Bron
  - Dijon
  - Lille
  - Paris
  - Saint-Herblain
  - Vénissieux
- Israel (5):
  - Holon
  - Jerusalem
  - Ofakim
  - Safed
  - Tel Litwinsky
- Italy (4):
  - Cinisello Balsamo
  - Napoli
  - Palermo
  - Roma
- Oslo (2 Locations), Norway
- United Kingdom (7):
  - Burton-on-Trent
  - Chesterfield
  - Isle of White
  - Londonderry/N. Ireland
  - Peterborough
  - Salford
  - Stevenage

REFERENCES:
- [Background] Moriarty PM, Jacobson TA, Bruckert E, Thompson PD, Guyton JR, Baccara-Dinet MT, Gipe D. Efficacy and safety of alirocumab, a monoclonal antibody to PCSK9, in statin-intolerant patients: design and rationale of ODYSSEY ALTERNATIVE, a randomized phase 3 trial. J Clin Lipidol. 2014 Nov-Dec;8(6):554-561. doi: 10.1016/j.jacl.2014.09.007. Epub 2014 Sep 19. PMID 25499937
- [Result] Moriarty PM, Thompson PD, Cannon CP, Guyton JR, Bergeron J, Zieve FJ, Bruckert E, Jacobson TA, Kopecky SL, Baccara-Dinet MT, Du Y, Pordy R, Gipe DA; ODYSSEY ALTERNATIVE Investigators. Efficacy and safety of alirocumab vs ezetimibe in statin-intolerant patients, with a statin rechallenge arm: The ODYSSEY ALTERNATIVE randomized trial. J Clin Lipidol. 2015 Nov-Dec;9(6):758-769. doi: 10.1016/j.jacl.2015.08.006. Epub 2015 Aug 29. PMID 26687696
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Moriarty PM, Thompson PD, Cannon CP, Guyton JR, Bergeron J, Zieve FJ, Bruckert E, Jacobson TA, Baccara-Dinet MT, Zhao J, Donahue S, Ali S, Manvelian G, Pordy R. Efficacy and safety of alirocumab in statin-intolerant patients over 3 years: open-label treatment period of the ODYSSEY ALTERNATIVE trial. J Clin Lipidol. 2020 Jan-Feb;14(1):88-97.e2. doi: 10.1016/j.jacl.2020.01.001. Epub 2020 Jan 13. PMID 32192644
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Defesche JC, Stefanutti C, Langslet G, Hopkins PN, Seiz W, Baccara-Dinet MT, Hamon SC, Banerjee P, Kastelein JJP. Efficacy of alirocumab in 1191 patients with a wide spectrum of mutations in genes causative for familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1338-1346.e7. doi: 10.1016/j.jacl.2017.08.016. Epub 2017 Sep 4. PMID 28964736
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 67 sites in 8 countries. Overall, 519 participants were screened between 28 September 2012 and 11 August 2013, 158 of whom were screen failures. Screen failures were mainly due to exclusion criteria met. After screening, 361 participants entered into a 4-week single blind placebo run-in period.
Pre-assignment Details: At the end of the single blind placebo run-in period, eligible participants were randomized to treatment arms centrally using a 2:2:1 (alirocumab:ezetimibe:atorvastatin) ratio. Randomization was stratified according to prior history of myocardial infarction or ischemic stroke. 314 participants were randomized.
Groups:
- Atorvastatin (Statin Rechallenge Arm): Atorvastatin 20 mg over-encapsulated tablets orally once daily (QD) for 24 weeks and placebo (for alirocumab) subcutaneous (SC) injection every two weeks (Q2W) for 24 weeks added to stable LMT.
- Ezetimibe (Active Comparator): Ezetimibe 10 mg over-encapsulated tablets orally QD for 24 weeks and placebo (for alirocumab) SC injection Q2W for 24 weeks added to stable LMT.
Period: Overall Study
Arm/Group | Atorvastatin (Statin Rechallenge Arm) | Ezetimibe (Active Comparator) | Alirocumab 75 mg/ up to 150 mg
Started | 63 | 125 | 126
Treated | 63 | 124 | 126
Completed | 42 | 82 | 96
Not Completed | 21 | 43 | 30
Not completed — Randomized but not treated | 0 | 1 | 0
Not completed — Adverse Event | 16 | 31 | 23
Not completed — Poor compliance to protocol | 2 | 0 | 0
Not completed — Other | 3 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin (Statin Rechallenge Arm): Atorvastatin 20 mg over-encapsulated tablets orally QD for 24 weeks and placebo (for alirocumab) SC injection Q2W for 24 weeks added to stable lipid-modifying therapy (LMT).
- Total: Total of all reporting groups
Arm/Group | Atorvastatin (Statin Rechallenge Arm) | Ezetimibe (Active Comparator) | Alirocumab 75 mg/ up to 150 mg | Total
Number analyzed (Participants) | 63 | 125 | 126 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.5) | 62.8 (10.1) | 64.1 (9.0) | 63.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 58 | 56 | 142
  Male | 35 | 67 | 70 | 172
Low Density Lipoprotein Cholesterol (LDL-C) in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C values were obtained from Friedewald formula.
  mg/dL | 187.3 (59.5) | 193.5 (70.9) | 191.1 (72.7) | 191.3 (69.3)
LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C values were obtained from Friedewald formula.
  mmol/L | 4.85 (1.54) | 5.011 (1.837) | 4.951 (1.883) | 4.954 (1.796)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent--To-Treat (ITT) Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -14.6 (2.2) | -45.0 (2.2)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Alirocumab group was compared to the corresponding active control group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -30.4, 95% CI 2-sided [-36.6 to -24.2]

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On--Treatment Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 118 | 123
percent change | -17.1 (2.0) | -52.2 (2.0)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 5% level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -35.1, 95% CI 2-sided [-40.7 to -29.5]

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL--C at Week 12 -- ITT Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -15.6 (2.0) | -47.0 (1.9)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -31.5, 95% CI 2-sided [-36.9 to -26.1]

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On--Treatment Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 12
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 118 | 123
percent change | -18.0 (1.8) | -51.2 (1.7)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -33.1, 95% CI 2-sided [-38.0 to -28.2]

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 -- ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post--baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 116 | 122
percent change | -11.2 (1.7) | -36.3 (1.7)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.1, 95% CI 2-sided [-29.8 to -20.4]

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 -- On--Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first).
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 95 | 109
percent change | -14.4 (1.4) | -42.6 (1.3)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -28.2, 95% CI 2-sided [-32.1 to -24.4]

7. Secondary Outcome: Percent Change From Baseline in Non--High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 -- ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -14.6 (1.7) | -40.2 (1.7)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.6, 95% CI 2-sided [-30.4 to -20.8]

8. Secondary Outcome: Percent Change From Baseline in Non--HDL-C at Week 24 -- On--Treatment Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the mITT population with one baseline and at least one post-baseline Non-HDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 118 | 123
percent change | -17.1 (1.5) | -46.9 (1.4)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -29.8, 95% CI 2-sided [-33.9 to -25.8]

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total--C) at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline total-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -10.9 (1.4) | -31.8 (1.4)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -20.8, 95% CI 2-sided [-24.7 to -17.0]

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 -- ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 116 | 122
percent change | -11.6 (1.5) | -36.1 (1.5)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -24.5, 95% CI 2-sided [-28.7 to -20.4]

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 12
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -15.8 (1.5) | -41.5 (1.5)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.7, 95% CI 2-sided [-29.9 to -21.5]

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 12
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Alirocumab 75/ up to 150: Alirocumab 75 mg SC injection Q2W for 24 weeks and placebo (for atorvastatin/ezetimibe) over-encapsulated tablets orally QD for 24 weeks added to stable LMT. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on cardiovascular risk.
Arm/Group | Ezetimibe | Alirocumab 75/ up to 150
Number analyzed (Participants) | 122 | 126
percent change | -11.6 (1.2) | -32.7 (1.2)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75/ up to 150; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -21.1, 95% CI 2-sided [-24.5 to -17.7]

13. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or Moderate or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from a multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included in the imputation model (ITT analysis).
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percentage of participants | 4.4 | 41.9
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant). Statistical analysis used a multiple imputation approach followed by a Logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 19.5, 95% CI 2-sided [6.9 to 55.2]

14. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or Moderate or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 were obtained from a multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 24 i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first (on-treatment analysis).
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 118 | 123
percentage of participants | 5.6 | 51.2
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 24.9, 95% CI 2-sided [8.6 to 71.9]

15. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: as for outcome 13
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percentage of participants | 0.8 | 32.5
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant). Statistical analysis used a last observation carried forward (LOCF) approach followed by Exact conditional logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Exact Conditional Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 71.5, 95% CI 2-sided [11.1 to 3022.1]

16. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: as for outcome 14
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 118 | 123
percentage of participants | 0.8 | 39.0
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant). Statistical analysis used a LOCF approach followed by Exact conditional logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Exact Conditional Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 109.8, 95% CI 2-sided [16.5 to 4759.3]

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 - ITT Analysis
Description: Combined Estimate for Adjusted Mean (Standard Error) at Week 24 from multiple imputation followed by robust regression including all available post-baseline data from Week 4 to Week 24 regardless of status on or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -7.3 (2.5) | -25.9 (2.4)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant). Statistical analysis used a multiple imputation approach followed by a robust regression model; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Adjusted Mean Difference = -18.7, 95% CI 2-sided [-25.5 to -11.8]

18. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | 6.8 (1.7) | 7.7 (1.7)
Statistical Analysis 1: Comparison: Ezetimibe vs Alirocumab 75 mg/ up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p = 0.6997, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 0.9, 95% CI 2-sided [-3.8 to 5.6]

19. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: as for outcome 17
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -3.6 (2.8) | -9.3 (2.7)

20. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 116 | 122
percent change | 2.9 (1.2) | 4.8 (1.2)

21. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12 -- ITT Analysis
Description: as for outcome 17
Time Frame: From Baseline to Week 12
Population: Lipoprotein(a) ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -4.5 (2.3) | -21.7 (2.2)

22. Secondary Outcome: Percent Change in HDL-C From Baseline to Week 12 -- ITT Analysis
Description: Least-squares (LS) means and standard errors (SE) taken from MMRM (mixed-effect model with repeated measures) analysis
Time Frame: From Baseline to Week 12
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | 7.6 (1.2) | 9.0 (1.2)

23. Secondary Outcome: Percent Change in Fasting Triglycerides From Baseline to Week 12 -- ITT Analysis
Description: as for outcome 17
Time Frame: From Baseline to Week 12
Population: Fasting Triglycerides ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 122 | 126
percent change | -9.4 (2.6) | -8.0 (2.5)

24. Secondary Outcome: Percent Change From Baseline in Apo A--1 at Week 12 -- ITT Analysis
Description: Least squares (LS) means and standard errors (SE) taken from MMRM (mixed effect model with repeated measures) analysis.
Time Frame: From Baseline to Week 12
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 116 | 122
percent change | 3.9 (1.0) | 5.5 (1.0)

25. Other Pre Specified Outcome: Percentage of Participants Who Experienced Skeletal Muscle-related Adverse Event (AE)
Description: Skeletal muscle-related adverse events were a predefined category including myalgia, muscle spasms, muscular weakness, musculoskeletal stiffness and muscle fatigue. Events that developed during treatment emergent adverse events period (the time from the first double-blindstudy treatment [injection or capsules, whichever came first] up to the day of the last double-blind injection + 70 days ) are reported.
Time Frame: From Baseline up to Week 24
Population: Safety population
Measure: Number; unit: Percentage of Participants
Groups:
- Atorvastatin (Statin Rechallenge Arm): Atorvastatin 20 mg over-encapsulated tablets orally QD for 24 weeks and placebo (for alirocumab) SC injection Q2W for 24 weeks added to stable LMT.
Arm/Group | Atorvastatin (Statin Rechallenge Arm) | Ezetimibe (Active Comparator) | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 63 | 124 | 126
Percentage of Participants
  Any skeletal muscle-related AE | 46.0 | 41.1 | 32.5
  Leading to treatment discontinuation | 22.2 | 20.2 | 15.9

26. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 Versus Atorvastatin - Raw Data Description - Intent-To-Treat (ITT) Analysis
Time Frame: From Baseline up to Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin (Statin Rechallenge Arm) | Ezetimibe (Active Comparator) | Alirocumab 75 mg/ up to 150 mg
Number analyzed (Participants) | 54 | 106 | 112
percent change | -31.9 (25.1) | -15.2 (22.4) | -47.3 (22.7)

ADVERSE EVENTS:
Time Frame: From Baseline up to the Last Double-Blind Injection Date + 70 Days
Description: Treatment emergent adverse events that developed during treatment emergent adverse events period (the time from the first double-blind study treatment [injection or capsules, whichever came first] up to the day of the last double-blind injection + 70 days ) are reported.
Groups:
- Atorvastatin: Atorvastatin 20 mg over-encapsulated tablets orally QD for 24 weeks and placebo (for alirocumab) SC injection Q2W for 22 weeks added to stable LMT.
- Ezetimibe: Ezetimibe 10 mg over-encapsulated tablets orally QD for 24 weeks and placebo for alirocumab SC injection Q2W for 22 weeks added to stable LMT.
- Alirocumab 75 mg/ up to 150 mg: Alirocumab 75 mg SC injection Q2W for 22 weeks and placebo for atorvastatin/ezetimibe over-encapsulated tablets orally QD for 24 weeks added to stable LMT. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL--C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on cardiovascular risk.
Arm/Group | Atorvastatin | Ezetimibe | Alirocumab 75 mg/ up to 150 mg
Serious Adverse Events (participants affected / at risk) | 7/63 | 10/124 | 12/126
Other Adverse Events (participants affected / at risk) | 35/63 | 63/124 | 57/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=63) | Ezetimibe (N=124) | Alirocumab 75 mg/ up to 150 mg (N=126)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Non-Cardiac chest pain (General disorders) | 1 | 4 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=63) | Ezetimibe (N=124) | Alirocumab 75 mg/ up to 150 mg (N=126)
Fatigue (General disorders) | 5 | 4 | 6
Nasopharyngitis (Infections and infestations) | 2 | 10 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 9 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 29 | 31
Headache (Nervous system disorders) | 4 | 6 | 6
Paraesthesia (Nervous system disorders) | 4 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.